CLINICAL TRIAL: NCT03584373
Title: Pain Outcomes of Non-opioid Analgesia After Ureteroscopy or Percutaneous Nephrolithotomy for Nephrolithiasis: a Prospective Randomized Controlled Trial.
Brief Title: Pain Outcomes of Non-opioid vs. Opioid Analgesia for Kidney Stone Surgery.
Acronym: PO-NOA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-9031
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Results first posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-10

CONDITIONS: Nephrolithiasis
Keywords: Pain Outcomes; Ureteroscopy; Percutaneous Nephrolithotomy; Opioids
MeSH Terms: conditions — Nephrolithiasis | interventions — Ketorolac; Ketorolac Tromethamine; Acetaminophen; oxycodone-acetaminophen

STUDY DESIGN:
Intervention Model Description: This will be an open label, prospective study of approximately 112 subjects undergoing either ureteroscopy or percutaneous nephrolithotomy. Patients who are eligible and choose to undergo ureteroscopy or percutaneous nephrolithotomy will then be asked if they would like to participate in the study and informed consent will be obtained. Patients will then be randomized to control (opioid analgesia) or non-opioid analgesia groups, and given this medication at discharge.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Non-Opioid Analgesia (Experimental): Ketorolac - Oral; 10 mg tablet: 1 tablet every 6 hours, or as needed. (20 tablets prescribed).
  Acetaminophen - Oral; patient directed as needed. Not prescribed.
  Ketorolac and Acetaminophen administered post surgery to compare pain outcomes to that of Percocet.
  Interventions: Drug: Ketorolac Oral Tablet [Toradol]; Drug: Acetaminophen
- Opioid Analgesia (Active Comparator): Percocet - Oral; 5 mg tablet: 1 tablet every 4-6 hours, or as needed. (10 tablets prescribed).
  Percocet administered post surgery to compare pain outcomes to that of the non-opioid analgesia.
  Interventions: Drug: Oxycodone Acetaminophen

INTERVENTIONS:
Drug: Ketorolac Oral Tablet [Toradol] — Ketorolac is a prescribed NSAID with strong analgesic activity. Ketorolac will be administered post surgery to compare pain outcomes to that of Percocet.
  Other Names: Toradol
  Arms: Non-Opioid Analgesia
Drug: Acetaminophen — Acetaminophen is an over-the counter pain medication that will be administered post surgery to compare pain outcomes to that of Percocet.
  Other Names: Tylenol
  Arms: Non-Opioid Analgesia
Drug: Oxycodone Acetaminophen — Percocet is a prescribed opioid medication to manage pain. Percocet will be administered post surgery to compare pain outcomes to that of non-opioid analgesia.
  Other Names: Percocet
  Arms: Opioid Analgesia

SUMMARY:
There are two options for postoperative pain management: opioid and non-opioid analgesia. Pain outcomes will be compared in patients undergoing ureteroscopy and percutaneous nephrolithotomy by randomly administering opioid and non-opioid analgesia.

DETAILED DESCRIPTION:
Perioperative pain is often managed by opioids. However, post surgical pain management with opioids can often lead to long-term opioid use; additionally, opioids can cause unwanted side effects including respiratory depression that can lead to hypoxia and respiratory arrest, as well as nausea, vomiting, pruritus, ileus, and constipation. As an alternative to opioid perioperative pain management, non-opioid analgesia has been proven to be as effective as opioid management in acute pain. Nonsteroidal Anti-inflammatory Drugs (NSAIDs) and acetaminophen are often utilized as alternatives to opioid analgesia, and have an increased efficacy when combined. Both NSAIDS and acetaminophen have been proven to decrease opioid requirements and have minimized opiate-induced adverse events.

In this randomized clinical trial, pain outcomes after ureteroscopy and percutaneous nephrolithotomy will be investigated in patients who are treated with opioids versus a non-opioid regimen of ketorolac and acetaminophen. Percutaneous nephrolithotomy and ureteroscopy are minimally invasive surgical techniques to surgically remove kidney stones. This trial will seek to determine whether non-opioid therapy is noninferior to opioid therapy in the determination of pain intensity as measured by an 11-point numeric rating scale, in which 0 indicates no pain and 10 indicates the worst possible pain, one week after the surgery by telephone call.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women age>18 years old
* Presence of renal or ureteral stones suitable for ureteroscopy or percutaneous nephrolithotomy.
* Uncomplicated ureteroscopy or percutaneous nephrolithotomy

Exclusion Criteria:

* Pregnant/Breastfeeding/Possibly Pregnant Patients
* Pediatric Patients
* Sensitive or Allergic to Opioids, Ketorolac, or Acetaminophen
* Significant Renal Disease
* Peptic Ulcer Disease
* Chronic Pain and recovering opiate use
* Inability to complete questionnaires
* Non-mobile patients
* Patients on methadone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara L Watts, MD, Principal Investigator — Montefiore
Locations (2):
- United States (2):
  - Jack D. Weiler Hospital, The Bronx, New York
  - Montefiore Hutchinson Campus, The Bronx, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients scheduled for surgery between July 2018 and May 2021 were consented and enrolled into the study.
Pre-assignment Details: A total of 119 patients were consented and enrolled into the study. Of the 119 patients, 14 patients screen failed (did not meet inclusion/exclusion criteria) and were not randomized into the study. Accordingly, 105 patients were randomized into the two arms/groups for this study.
Groups:
- Non-Opioid Analgesia: Ketorolac - Oral; 10 mg tablet: 1 tablet every 6 hours, or as needed. (20 tablets prescribed).
  Acetaminophen - Oral; patient directed as needed. Not prescribed.
  Ketorolac and Acetaminophen administered post surgery to compare pain outcomes to that of Percocet.
  Ketorolac Oral Tablet [Toradol]: Ketorolac is a prescribed NSAID with strong analgesic activity. Ketorolac will be administered post surgery to compare pain outcomes to that of Percocet.
  Acetaminophen: Acetaminophen is an over-the counter pain medication that will be administered post surgery to compare pain outcomes to that of Percocet.
- Opioid Analgesia: Percocet - Oral; 5 mg tablet: 1 tablet every 4-6 hours, or as needed. (10 tablets prescribed).
  Percocet administered post surgery to compare pain outcomes to that of the non-opioid analgesia.
  Oxycodone Acetaminophen: Percocet is a prescribed opioid medication to manage pain. Percocet will be administered post surgery to compare pain outcomes to that of non-opioid analgesia.
Period: Overall Study
Arm/Group | Non-Opioid Analgesia | Opioid Analgesia
Started | 51 | 54
Completed | 44 | 46
Not Completed | 7 | 8
Not completed — Lost to Follow-up | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Opioid Analgesia | Opioid Analgesia | Total
Number analyzed (Participants) | 51 | 54 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (15.8) | 47 (14.7) | 48 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 54
  Male | 24 | 27 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 5 | 3 | 8
  Non-Hispanic Black | 8 | 10 | 18
  Hispanic | 22 | 33 | 55
  Other/Unknown | 16 | 8 | 24
Region of Enrollment [Number; unit: participants]
  United States | 51 | 54 | 105
Body Mass Index (BMI) [Median (Standard Deviation); unit: kg/m^2] | 29.0 (5.8) | 29.2 (6.3) | 29.1 (6.0)
Participants with Percutaneous Nephrolithotomy (PCNL) Surgeries [Count of Participants; unit: Participants] | 13 | 18 | 31
Stent Placement During Procedure [Count of Participants; unit: Participants] | 33 | 35 | 68
Prior Kidney Stone Removal Surgery [Count of Participants; unit: Participants] | 23 | 15 | 38
Average Stone Burden [Mean (Standard Deviation); unit: millimeters] | 10.9 (4.5) | 18.1 (12.1) | 14.7 (9.8)

OUTCOME MEASURES:

1. Primary Outcome: Satisfaction With Pain Relief
Description: The patient will be administered a survey and asked to rate satisfaction with pain relief since the time of surgery and being on the assigned medication. Scoring will be on an 11-point ordinal numeric rating scale, with 0 being not satisfied with pain relief, and 10 being well-satisfied. Higher scores are indicative of greater satisfaction with pain relief
Time Frame: 1 week post surgery
Population: Data was not collected and analyzed for the 7 participants who were lost to follow up in the non-opioid analgesia arm and 8 participants who were lost to follow up in the opioid analgesia arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Opioid Analgesia | Opioid Analgesia
Number analyzed (Participants) | 44 | 46
score on a scale | 8.70 (2.01) | 8.85 (1.49)
Statistical Analysis 1: Comparison: Non-Opioid Analgesia vs Opioid Analgesia; Test type: Non-Inferiority — Non-inferiority margin of 1.3; p = 0.70, t-test, 2 sided; Mean Difference (Net) = -0.14, 95% CI 2-sided [-0.89 to 0.60]

2. Primary Outcome: Current Pain Intensity Level
Description: The patient will be administered a survey and asked to rate their current pain intensity level (1 week post surgery) on an 11-point ordinal numeric rating scale ranging from 0-10, with 0 being no pain, and 10 being the worst possible pain. Higher scores are indicative of greater pain intensity.
Time Frame: 1 week post surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Opioid Analgesia | Opioid Analgesia
Number analyzed (Participants) | 44 | 46
score on a scale | 1.14 (1.94) | 1.37 (2.08)
Statistical Analysis 1: Comparison: Non-Opioid Analgesia vs Opioid Analgesia; Test type: Non-Inferiority — Non-inferiority margin of 1.3; p = 0.58, t-test, 2 sided; Mean Difference (Net) = -0.23, 95% CI 2-sided [-1.08 to 0.61]

3. Primary Outcome: Peak Pain Intensity Level
Description: The patient will be administered a survey and asked to rate the worst/peak pain intensity level since undergoing the surgery. The patient will be asked to rate this worst pain intensity level on an 11-point ordinal numeric rating scale ranging from 0-10, with 0 being no pain, and 10 being the worst possible pain. Higher scoring is indicative of worst/peak pain intensity level since the time of surgery
Time Frame: 1 week post surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Opioid Analgesia | Opioid Analgesia
Number analyzed (Participants) | 44 | 46
score on a scale | 5.61 (3.41) | 7.52 (3.00)
Statistical Analysis 1: Comparison: Non-Opioid Analgesia vs Opioid Analgesia; Test type: Non-Inferiority — Non-inferiority margin of 1.3; p = 0.006, t-test, 2 sided; Mean Difference (Net) = -1.91, 95% CI 2-sided [-3.25 to -0.56]

4. Primary Outcome: Average Pain Intensity Level
Description: The patient will be administered a survey and asked to rate their average pain intensity level since undergoing surgery. The patient will be asked to rate this average pain intensity level on an 11-point ordinal numeric rating scale ranging from 0-10, with 0 being no pain, and 10 being the worst possible pain. Higher scores are indicative of higher average pain intensity.
Time Frame: 1 week post surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Opioid Analgesia | Opioid Analgesia
Number analyzed (Participants) | 44 | 46
score on a scale | 3.34 (2.57) | 4.50 (2.69)
Statistical Analysis 1: Comparison: Non-Opioid Analgesia vs Opioid Analgesia; Test type: Non-Inferiority — Non-inferiority margin of 1.3; p = 0.04, t-test, 2 sided; Mean Difference (Net) = -1.16, 95% CI 2-sided [-2.26 to -0.06]

5. Primary Outcome: Perception of an Acceptable Pain Intensity Level
Description: The patient will be administered a survey and asked to rate what their perception or belief of an acceptable pain intensity level would be since undergoing the surgery. The patient will be asked to rate this acceptable pain intensity level on an 11-point ordinal numeric rating scale ranging from 0-10, with 0 equaling no pain, and 10 being the worst possible pain. Higher scores are indicative of the patient's belief of an acceptable pain intensity level.
Time Frame: 1 week post surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Opioid Analgesia | Opioid Analgesia
Number analyzed (Participants) | 44 | 46
score on a scale | 2.73 (2.48) | 3.28 (2.85)
Statistical Analysis 1: Comparison: Non-Opioid Analgesia vs Opioid Analgesia; Test type: Non-Inferiority — Non-inferiority margin of 1.3; p = 0.33, t-test, 2 sided; Mean Difference (Net) = -0.55, 95% CI 2-sided [-1.67 to 0.56]

6. Secondary Outcome: Unused Medications - Proportion of Prescribed Pills Unused at 1 Week Post-Surgery
Description: Unused medications is defined as the proportion of prescribed pills that were unused at 1 week post surgery as reported by the patient. More unused medications may indicate the potential to decrease the dosage needed.
Time Frame: 1 week post surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: proportion of unused pills
Arm/Group | Non-Opioid Analgesia | Opioid Analgesia
Number analyzed (Participants) | 44 | 46
proportion of unused pills | 0.63 (0.37) | 0.58 (0.35)
Statistical Analysis 1: Comparison: Non-Opioid Analgesia vs Opioid Analgesia; Test type: Non-Inferiority — Non-inferiority margin of 1.3; p = 0.47, t-test, 2 sided; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.10 to 0.21]

7. Secondary Outcome: Rates of Constipation
Description: Percentage of patients who experienced constipation any time during the week after surgery. A lower percentage of constipation may indicate less incidence of adverse events.
Time Frame: 1 week post surgery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Non-Opioid Analgesia | Opioid Analgesia
Number analyzed (Participants) | 44 | 46
Participants | 11 | 17

ADVERSE EVENTS:
Time Frame: Up to 1 week postoperatively
Arm/Group | Non-Opioid Analgesia | Opioid Analgesia
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/54
Serious Adverse Events (participants affected / at risk) | 5/51 | 7/54
Other Adverse Events (participants affected / at risk) | 2/51 | 1/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Opioid Analgesia (N=51) | Opioid Analgesia (N=54)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2) — Verbatim, Dysuria or Pain with Urination
Anemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Verbatim, epigastric and lower left quadrant pain
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Verbatim, bowel movements
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-Opioid Analgesia (N=51) | Opioid Analgesia (N=54)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) — Secondary to Anemia
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT03584373/Prot_SAP_000.pdf